CLINICAL TRIAL: NCT01109394
Title: Comprehensive Omics Analysis of Pediatric and Adult Solid Tumors and Establishment of a Repository for Related Biological Studies
Status: Recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 100086; 10-C-0086
Record Dates: First submitted 2010-04-22; First posted 2010-04-23 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2025-09-25

CONDITIONS: Sarcoma; Endocrine Tumors; Neuroblastoma; Retinoblastoma; Renal Cancer
Keywords: Genomics; Proteomics; Tissue Repository; Omics; Cell Lines; Natural History; Pediatric Cancer; Solid Tumor; Sarcoma; Kidney Cancer; Neuroblastoma
MeSH Terms: conditions — Sarcoma; Neuroblastoma; Retinoblastoma; Kidney Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 1/Cohort 1: Adult or Pediatric subjects, with any malignancy, pre-malignancy, suspected malignancy, family history of malignancy, or without malignancy undergoing surgery or well visit.
- 2/Cohort 2: Human samples, specimens and data collected on IRB approved protocols that are now closed
- 3/Cohort 3: Parent/caregiver of a participating pediatric or adult subject who is being treated for, or who has previously been treated for any form of pediatric cancer.

SUMMARY:
Background:

- Laboratory investigators who are studying common childhood cancers are interested in developing a tissue repository to collect and store blood, serum, tissue, urine, or tumors of children who have cancer or adults who have common childhood cancers. To develop this repository, additional samples will be collected from children and adults who have been diagnosed with common childhood cancers such as leukemia and tumors of the central nervous system.

Objectives:

- To collect and store blood, serum, tissue, urine, or tumor samples of children who have cancer or adults who have common childhood cancers.

Eligibility:

* Individuals who have been diagnosed with a common childhood cancer (e.g., leukemia) regardless of patient age.
* Children, adolescents, and adults who have been diagnosed with a type of cancer more commonly found in adults.

Design:

* Extra blood, serum (the liquid part of blood), tissue, urine, or tumor samples will be collected from participants at a time when sampling is required for medical care or as part of a research study.
* No additional procedures will be performed for the sole purpose of obtaining additional tumor tissue, aside from what is required for clinical care.

DETAILED DESCRIPTION:
Background:

-Laboratory-based investigations have contributed to an improved understanding of the biology of cancer and to the development of new therapies for pediatric malignancies.

Objectives:

-Systematic Molecular, Genomic, Proteomic, Metabolomic ("Omic") and other profiling for enrolled subjects where omics refers to mechanistic studies using a set of advanced technologies to capture comprehensive aspects of biological systems providing insights into structure, function and interactions to understand these complex processes and diseases better.

Eligibility:

Pediatric or Adult subjects of any age with one of the following:

* Diagnosis of any tumor or malignancy, pre-malignant disorder or suspected cancer susceptibility familial syndromes, regardless of age
* Individuals without malignancy undergoing surgery, other treatment such as apheresis or normal well visit or routine blood draw as part of standard of care.
* Biological relatives of a subject with a tumor or malignancy (pediatric or adult) or with suspected familial cancer syndrome. Patients enrolled in an approved companion protocol
* Blood and/or tissue specimens that have been previously collected and are available for research analysis
* Biospecimens can be collected with minimal additional risk to the subject during sampling or procedures required for routine patient care.

Design:

* This study will allow for the collection of specimens for a Tissue Repository, and for designated sample investigations including systematic molecular, genomic and proteomic (Omic) profiling, and growth factor and cellular profile investigations.
* Testing activities may include:

  * DNA, RNA and protein extracted from a section of tumor and normal samples; the remainder will be stored.
  * Germ line DNA and RNA extracted from lymphocytes or other normal uninvolved tissue
  * Germ line DNA will be extracted from lymphocytes or other normal uninvolved tissue of relatives of the subject.
  * Xenografts, explant and cell lines established from tumor, pre-malignant and normal samples
  * Tumor samples and samples for circulating tumor cells sent for the establishment of Xenografts and single cell suspension of tumor for drug testing or for monitoring cell free DNA over time
  * Omics (Genomics and Proteomic) studies will be performed
  * Growth factor and cellular profile investigations of bone marrow-derived cell populations to include quantification of hematopoietic progenitor cells (HPCs), endothelial progenitor cells (EPCs), and mesenchymal progenitor cells (MPCs), levels of matrix metalloprotease 2 and 9 (MMP2) and (MMP9), gene expression, growth factor and microvesicle analysis and bone marrow analysis of progenitor cells in blood and tissue.
  * Research tests described in active IRB approved protocols.
  * Immune profiling and stromal profiling of blood, tumor, and normal tissues
  * Immune function studies from blood and normal tumor tissues.
* Utilizing an oversight committee to oversee the receipt and the distribution of unlinked tissues to other investigators.
* Qualitative methodologies will be used to ascertain knowledge, attitudes, beliefs, and behaviors in 25-35 parents/caregivers at NIH concerning the anticipated use of NGS for diagnosing and directing therapy for pediatric cancer and how incidental findings might be returned.
* Expected accrual of 100-150 patients per year.

ELIGIBILITY:
* SUBJECT INCLUSION CRITERIA:

Pediatric or adult subjects with one of the following:

* Diagnosis of any tumor, malignancy, pre-malignant disorder, or suspected premalignant familial syndromes, regardless, of patient age;
* Biological relatives of any patient with a tumor, malignancy, pre-malignant disorder, or suspected familial pre-malignant syndrome, regardless of patient age or the diagnosis of an adult malignancy or pre-malignant disorder;
* Healthy Volunteer without history of malignancy nor a family member currently being treated for cancer who are undergoing surgery, treatment or during well visits;
* Biospecimens can be collected with minimal additional risk to the subject during sampling or procedures required for routine patient care.
* Human samples, specimens and data collected on IRB approved protocols that are now closed
* Ability of subject, Legally Authorized Representative (LAR), or parent/legal guardian of children <=18 to understand and be willing to sign an IRB-approved informed consent document that permits the use of the tumor and other samples for genomic-based molecular characterization projects.

Inclusion Criteria for Social and Behavioral Outcome Interviews:

* Parent/caregiver of a participating pediatric or adult patient who is being treated for, or who has previously been treated for any form of pediatric cancer.
* Must be able to give consent and sign the informed consent document.
* Able to understand the English language.

EXCLUSION CRITERIA:

None

Min Age: 4 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with a diagnosis of any tumor or malignancy regardless of age, or without malignancy undergoing surgery, other treatment or normal well visit. Suspicion of a familial premalignant condition. Biological relatives of a subject with a pediatric or adult tumor or malignancy or with suspected familial cancer syndrome.
Sampling Method: Non-Probability Sample
Enrollment: 6035 (Estimated)
Dates: Start 2010-04-21 (Actual)

PRIMARY OUTCOMES:
tissue analysis | ongoing
  Perform systematic molecular, genomic, proteomic, metabolomics and other high throughput ( Omics ) profiling on tumor and normal tissues

CONTACTS AND LOCATIONS:
Overall Officials: Rosandra N Kaplan, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (5):
- United States (5):
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Hospital of Orange County (CHOC Children's), Orange, Florida
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Tisch Cancer Institute, Mount Sinai Medical Center, New York, New York
  - Carolinas Medical Center/Levine Children's Hospital, Charlotte, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely. Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI. Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- [Background] Linet MS, Ries LA, Smith MA, Tarone RE, Devesa SS. Cancer surveillance series: recent trends in childhood cancer incidence and mortality in the United States. J Natl Cancer Inst. 1999 Jun 16;91(12):1051-8. doi: 10.1093/jnci/91.12.1051. PMID 10379968
- [Background] Khan J, Bittner ML, Chen Y, Meltzer PS, Trent JM. DNA microarray technology: the anticipated impact on the study of human disease. Biochim Biophys Acta. 1999 Mar 25;1423(2):M17-28. doi: 10.1016/s0304-419x(99)00004-9. PMID 10214349
- [Background] Khan J, Saal LH, Bittner ML, Chen Y, Trent JM, Meltzer PS. Expression profiling in cancer using cDNA microarrays. Electrophoresis. 1999 Feb;20(2):223-9. doi: 10.1002/(SICI)1522-2683(19990201)20:23.0.CO;2-A. PMID 10197427
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2010-C-0086.html